CLINICAL TRIAL: NCT03158324
Title: Phase IIa Dose-Expansion and Biomarker Study of OPB-111077 in An Enriched Population of Treatment-Refractory Advanced Solid Tumors
Brief Title: Phase IIa Dose-Expansion and Biomarker Study of OPB-111077
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/01181
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-04

CONDITIONS: NPC; Refractory Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Two parallel cohorts will be implemented: i. patients with tumors predicted to be dependent on oxidative phosphorylation metabolism or oncogene addicted tumors which have developed resistance to primary TKI therapy, or ii. patients with nasopharyngeal carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced refractory solid tumors (Experimental): Patients with advanced refractory solid tumors will be enrolled.
  Interventions: Drug: OPB-111077

INTERVENTIONS:
Drug: OPB-111077 — Receive 600 mg of OPB-111077 on a 4 days-on, 3 days-off per week in 28-day cycles till disease progression or intolerable toxicity

SUMMARY:
This is a phase IIa open-label, non-randomized dose-expansion study of OPB-111077 in patients with advanced, treatment refractory cancers who have biopsy-amenable lesions at study entry.

DETAILED DESCRIPTION:
This is a phase IIa open-label, non-randomized dose-expansion study of OPB-111077 in patients with advanced, treatment refractory cancers who have biopsy-amenable lesions at study entry. Patients on the proposed study will be treated with the RPII dose of OPB-111077 (600mg on a 4 days-on, 3 days-off per week schedule). They will be enrolled in two parallel cohorts: i. patients with tumors predicted to be dependent on oxidative phosphorylation metabolism or oncogene addicted tumors which have developed resistance to primary TKI therapy, or ii. patients with nasopharyngeal carcinoma

Each cohort will contain 11-26 patients, over a period of 12-36 months. Subjects will receive OPB-111077 in 28-day cycles till disease progression or intolerable toxicity. Mandatory tumour biopsies will be performed at baseline and on cycle 1 day 15 (where feasible and accessible). Circulating biomarker blood sampling will be performed on days 1, 11 and 15 of cycle 1, and upon completion of OPB-111077 dosing. Pharmacokinetics blood sampling will be performed on days 11 and 15 of cycle 1. Safety assessments will be performed on cycle 1 day 1, cycle 1 day 8, cycle 1 day 15, bi-weekly till week 8, then monthly thereafter and response assessments will be performed every 8 weeks. Metabolic response assessment by PET/CT will be performed after 2 cycles of treatment, while radiologic response assessment will be performed after every 2 cycles of OPB-111077 from cycle 4 onwards.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, locally recurrent or metastatic solid tumors, who have failed standard treatment
2. Subjects with NPC will be eligible as long as they have received prior platinum therapy
3. Subjects with other types of solid tumors will be eligible if: i) their archival tumor sample shows over-expression oxidative phosphorylation markers e.g., PGC-1α/ SIRT1 or ii) they have oncogene-addicted cancers (e.g., EGFR mutation-positive NSCLC, EML4-ALK fusion NSCLC, BRAF-mutant melanomas, GIST, RET-driven thyroid cancers) which have become resistant to primary TKI therapy
4. All subjects must have at least one tumour lesion (primary or metastatic) that is suitable for free-hand or image-guided biopsy at baseline.
5. Age ≥ 21 years, Eastern Cooperative Oncology Group (ECOG) performance status < 1
6. Adequate bone marrow, liver and renal function
7. Baseline serum lactate ¬<3mmol/l
8. Capable of swallowing tablets
9. Recovery from any previous drug- or procedure-related toxicity to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 Grade 0 or 1 (except alopecia), or to baseline preceding the prior treatment.
10. Signed informed consent obtained before any study specific procedure. Subjects must be able to understand and be willing to sign the written informed consent.

Exclusion Criteria:

1. Chemotherapy, radiotherapy, surgery, immunotherapy or other therapy within 3 weeks of starting investigational medicinal product (IMP).
2. Use of any prohibited medications (CYP3A4 inhibitors and inducers) or medications which may predispose to lactic acidosis (e.g., metformin, nucleoside analogue reverse within 1 week prior to start of study drug administration
3. Pregnancy or breastfeeding.
4. Women of childbearing potential not employing adequate contraception. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of study medication, and a negative result must be documented before start of study medication. Women of childbearing potential and men, must agree to use adequate contraception (barrier method of birth control) upon signing the informed consent form until at least 3 months after the last study drug administration.
5. Known or suspected allergy to the investigational agent or any agent given in association with this study.
6. Concurrent cancer which is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumours (Ta, Tis & T1) or any cancer curatively treated less than 3 years prior to study entry.
7. Interstitial lung disease with ongoing signs and symptoms at the time of screening.
8. Patients with CTCAE Grade 2 or higher peripheral neuropathy.
9. History of significant cardiac disease: congestive cardiac failure > NYHA class II, ongoing unstable angina, new-onset angina or myocardial infarction within the past 3 months

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-05-22 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rates | 3 years
  This will be calculated as the percentage of evaluable patients achieving complete and partial response with OPB-111077 treatment, according to the RECIST 1.1 criteria

SECONDARY OUTCOMES:
Metabolic response rates | 3 years
  This will be calculated as the percentage of evaluable patients achieving complete and partial metabolic response on 18F]-FDG PET/CT after 2 cycles of OPB-111077, as determined by the EORTC PET response criteria.
Progression free survival | 3 years
  This is defined as the time from the start of study treatment to documented progression of disease or death.
Haematologic and non-haematologic toxicities (all grades) | 3 years
  To evaluate the haematologic and non-haematologic toxicities of OPB-111077

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam MM, Lal S, FitzGerald KE, Zhang L. A holistic view of cancer bioenergetics: mitochondrial function and respiration play fundamental roles in the development and progression of diverse tumors. Clin Transl Med. 2016 Mar;5(1):3. doi: 10.1186/s40169-016-0082-9. Epub 2016 Jan 26. PMID 26812134
- [Background] Vellinga TT, Borovski T, de Boer VC, Fatrai S, van Schelven S, Trumpi K, Verheem A, Snoeren N, Emmink BL, Koster J, Rinkes IH, Kranenburg O. SIRT1/PGC1alpha-Dependent Increase in Oxidative Phosphorylation Supports Chemotherapy Resistance of Colon Cancer. Clin Cancer Res. 2015 Jun 15;21(12):2870-9. doi: 10.1158/1078-0432.CCR-14-2290. Epub 2015 Mar 16. PMID 25779952